CLINICAL TRIAL: NCT03390855
Title: Effects of the Consumption of Broccoli Sprouts in Overweight Subjects
Acronym: SPROUTvsFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Collaborators: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Débora Villaño, Proffesor, Universidad Católica San Antonio de Murcia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AGL-2013-46247-P
Record Dates: First submitted 2017-12-28; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Inflammation
Keywords: IL-6; Glucosinolate; Brassica oleracea; Sulphoraphane; Biomarkers; Bioavailability; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Intervention Model Description: The intervention consisted on a 10-week period which included daily consumption of a portion (30 g) of raw, fresh broccoli sprouts. After the intervention period, a follow-up recovery period for all subjects continued for other 90 days with no ingestion of broccoli sprouts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Broccoli sprout and follow up (Experimental): Daily consumption of 30 g of raw, fresh, broccoli sprouts, not cooked, during 10 weeks (70 days), followed by other 90 days of no ingestion of broccoli sprouts
  Interventions: Other: Broccoli sprouts

INTERVENTIONS:
Other: Broccoli sprouts

SUMMARY:
Nowadays there is an increasing demand by consumers on healthy food products prepared in convenient forms, simple to use and not containing additives. In this sense, broccoli sprouts (Brassica oleraceae var. italica) represent an interesting choice as they are rich in glucosinolates, nitrogen-sulfur compounds, that are believed to counteract the negative effects of diverse pathologies.

Human studies have been focused on the antitumoral properties of these vegetables, however there is less evidence on the anti-inflammatory properties of cruciferous vegetables in humans.

As obesity is linked to an inflammatory component, the aim of the study is to evaluate the anti-inflammatory action of broccoli sprouts in overweight adult subjects.

DETAILED DESCRIPTION:
We performed an interventional follow-up study to evaluate the effect of the daily consumption of broccoli sprouts during 10 weeks (70 days). The study was conducted at the Catholic University of Murcia under supervision of Consejo Superior de Investigaciones Científicas (CSIC).

The study was performed according with the Helsinki Declaration of Human Studies and approved by the Ethical Committee of the Catholic University of Murcia as well as the Bioethics Sub-Committee of the CSIC' Department of Ethics for the AGL-2013-46247-P project. Volunteers (n=40; 21 M, 19 W) were recruited in the Catholic University of Murcia (UCAM) and all of them were informed on the characteristics of the study and they signed the written-informed consent. Dietetic and life style habits were recorded from all participants. There were no drop-outs during the whole period of study and no adverse effects were reported due to the broccoli sprout ingestion.

One week before the beginning of the intervention period, subjects were asked to avoid the consumption of Brassica vegetables (broccoli, radish, cauliflower, Brussel sprouts, mustards, among others) and their derived products, and to follow a well-balanced diet (based on Mediterranean diet), with no other food restriction criteria. These dietary instructions were maintained during the entire period of study. Besides, they were requested to record any sign of adverse effect, illness or deviation of the experimental diet. The subjects maintained their usual lifestyles during the study.

On the first day, participants were given the portions of fresh broccoli sprouts to be taken for the whole week (7 trays of broccoli sprouts of 30 g each) and each week they had an appointment to provide them the fresh products. The intervention consisted on a 10-week period which included daily consumption of a portion (30 g) of raw, fresh broccoli sprouts. This amount is consistent with a half- serving according to WHO. Subjects were instructed to ingest 1 tray per day and to keep the trays refrigerated (4º C) at home. The intake of the broccoli sprouts was included in their normal daily diet and no specific time of consumption was established, with the only limitation of avoid cooking of the sprouts and to consume them fresh. Cooking procedures can affect the content of glucosinolates as well as their bioavailability and therefore some recipes were provided to the participants to facilitate the intake of the sprouts without affecting the phytochemical composition and absorption. After the intervention period, a follow-up recovery period for all subjects continued for other 90 days with no ingestion of broccoli sprouts.

Fasting blood samples and 24-h urine samples were taken on day 0 (jst before starting the intervention), day70 (end of intervention period), day 90 (20 days after end of intervention) and day 160 (90 days after end of intervention). Blood samples were collected from each subject by venipuncture from the antecubital vein; 3 mL were placed in heparin tubes and centrifuged at 10000 rpm for 10 min at 4ºC. Plasma was aliquoted and stored at -80ºC until analysis. Analysis were performed once each period was finished and in the same batch to minimize analytical variations. The total volume of the 24h-urine was recorded to calculate the absolute amounts of the compounds and metabolites excreted in the study period and aliquots were frozen at -80ºC for further analysis. Body weight and percentage of fat mass were measured as well and BMI calculated in each sampling time point.

Markers of inflammation as IL-6, C-reactive protein, IL-1β and TNF-α in plasma were determined in our laboratory using high-sensitivity ELISA kits.

Levels of glucosinolates, isothiocyanates and their metabolites were measured in urine by a rapid, sensitive and high throughput UHPLC-QqQ-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

BMI within the overweight range according to the World Health Organization criteria (24.9-29.9 kg/m2), aged 35-55 years, taking no vitamins, supplements or medication during the previous two months; no-smoking.

Exclusion Criteria:

Diagnosed diseases as hypertension and cardiovascular pathologies, diabetes, hepatic, gastrointestinal and renal diseases, as well as the intake of drugs related to these pathologies, vegetarian diet, pregnancy or breastfeeding.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in IL-6 levels | Changes observed from baseline at day 0 compared to 70, 90, 160 days
  Plasma levels of IL-6 measured at days 0, 70, 90 and 160 days of intervention
Change in C-reactive protein | Changes observed from baseline at day 0 compared to 70, 90, 160 days
  Plasma levels of C-reactive protein measured at days 0, 70, 90 and 160 days of intervention

SECONDARY OUTCOMES:
Bioavailability of glucosinolates from broccoli sprouts | Changes observed from baseline at day 0 compared to 70, 90, 160 days
  24 h-urine levels of glucosinolates and their metabolites measured by UHPLC-MS/MS

CONTACTS AND LOCATIONS:
Overall Officials: Diego Ángel Moreno Fernández, PhD, Principal Investigator — National Research Council, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baenas N, Villano D, Garcia-Viguera C, Moreno DA. Optimizing elicitation and seed priming to enrich broccoli and radish sprouts in glucosinolates. Food Chem. 2016 Aug 1;204:314-319. doi: 10.1016/j.foodchem.2016.02.144. Epub 2016 Feb 26. PMID 26988507
- [Background] Baenas N, Suarez-Martinez C, Garcia-Viguera C, Moreno DA. Bioavailability and new biomarkers of cruciferous sprouts consumption. Food Res Int. 2017 Oct;100(Pt 1):497-503. doi: 10.1016/j.foodres.2017.07.049. Epub 2017 Jul 21. PMID 28873713
- [Derived] Lopez-Chillon MT, Carazo-Diaz C, Prieto-Merino D, Zafrilla P, Moreno DA, Villano D. Effects of long-term consumption of broccoli sprouts on inflammatory markers in overweight subjects. Clin Nutr. 2019 Apr;38(2):745-752. doi: 10.1016/j.clnu.2018.03.006. Epub 2018 Mar 13. PMID 29573889